CLINICAL TRIAL: NCT01896908
Title: Effect of Dietary Sodium Restriction in the Management of Patients With Heart Failure and Preserved Ejection Fraction: a Randomized Clinical Trial
Brief Title: Effect of Dietary Sodium Restriction in the Management of Patients With Heart Failure and Diastolic Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HCPA - 120437
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-08

CONDITIONS: Diastolic Dysfunction
Keywords: diastolic dysfunction; Sodium restriction; Randomized clinical trial

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Sodium restriction (1.6g sodium daily - 4g salt) combined with 800 ml of fluid intake
  Interventions: Other: Sodium restriction
- Control (No Intervention): Normal sodium diet (4g sodium daily - 10g salt) and free fluid intake

INTERVENTIONS:
Other: Sodium restriction — Patients that are eligible and fulfill the inclusion criteria will be invited to participate while hospitalized, and then sign the informed consent form. Then, the dietitian on call will be notified in order to change the dietary map of the patients. The prescription diet for both the intervention and control group will be the same: DIET AS RESEARCH PROTOCOL. PATIENT WILL RECEIVE THE DIET UNTIL DAY __ / __ OR DISCHARGE. PLEASE DO NOT CHANGE IT. This will be combined with the medical staff and with the Nutrition and Dietetics service.
  The evaluation of outcomes after hospital discharge will be held in the institution of reference when will be performed clinical evaluation and blood samples collection for neurohormonal activation analysis.
  Arms: Intervention

SUMMARY:
Although half of the patients with HF has normal ejection fraction or slightly altered (HF-PEF) and the prognosis differs little from those with reduced ejection fraction, the pathophysiology of HF-PEF is still poorly understood.

Sodium restriction is the most common measure of self-care oriented to HF patients for management of congestive episodes. The role of this orientation in the treatment of patients with preserved ejection fraction, however, is still unclear. The evaluation of the effects of sodium restriction on neurohormonal activation and episodes of decompensation in HF-PEF can promote a better understanding of the pathophysiological progression of this complex syndrome.

DETAILED DESCRIPTION:
This is a randomized, parallel trial with blinded outcome assessment. The sample will include adult patients (aged ≥18 years) with a diagnosis of HF-PEF admitted for HF decompensation. The patients will be randomized to receive a diet with sodium and fluid intake restricted to 0.8 g/day and 800 mL/day respectively (intervention group) or an unrestricted diet, with 4 g/day sodium and unlimited fluid intake (control group), and followed for 7 days or until hospital discharge. The primary outcome shall consist of weight loss at 7 days or discharge. The secondary outcome includes assessment of clinical stability, neurohormonal activation, daily perception of thirst and readmission rate at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes
* Age equal to or above 18 years
* Diagnosis of heart failure whit preserved ejection fraction (LVEF> 50%)
* Patients hospitalized for heart failure decompensation whit hospital admission within 36 hours, who agree to participate in the study by signing the informed consent.

Exclusion Criteria:

* Patients who present values of endogenous creatinine clearance less than or equal to 30 ml / min;
* Cardiogenic shock,
* Those with survival compromised by another disease in evolution and / or difficulty adhering to treatment (dementia, cognitive impairment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2016-07-31 (Actual)

PRIMARY OUTCOMES:
Weight loss | seven days or hospital discharge

SECONDARY OUTCOMES:
Assessment of clinical stability | Seven days or hospital discharge
  Symptomatic improvement without evidence of congestion (congestion score)
  Weight stable for two days, without changing more than 1kg, (daily weight)
  Without IV drug for HF for 48 hours (daily record of medication: diuretics, vasodilators)
  No increase in diuretic dose for 48 hours (daily records of medications)
Neurohormonal activation | On admission and at discharge
  Assessment of neurohormonal activation shall include measurement of serum renin, aldosterone, and BNP levels.
Daily perception of thirst | Seven days or hospital discharge
  A visual scale (with values ranging from 0 to 10) will be used daily to verify the degree of thirst.
Readmission rate at 30 days | Patients shall be followed for 30 days after discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Eneida Rabelo da Silva, ScD, Principal Investigator — HCPA
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Machado d'Almeida KS, Rabelo-Silva ER, Souza GC, Trojahn MM, Santin Barilli SL, Aliti G, Rohde LE, Biolo A, Beck-da-Silva L. Aggressive fluid and sodium restriction in decompensated heart failure with preserved ejection fraction: Results from a randomized clinical trial. Nutrition. 2018 Oct;54:111-117. doi: 10.1016/j.nut.2018.02.007. Epub 2018 Mar 21. PMID 29793053
- [Derived] d'Almeida KS, Rabelo-Silva ER, Souza GC, Trojahn MM, Barilli SL, Mansson JV, Biolo A, Rohde LE, Clausell N, Beck-da-Silva L. Effect of fluid and dietary sodium restriction in the management of patients with heart failure and preserved ejection fraction: study protocol for a randomized controlled trial. Trials. 2014 Sep 4;15:347. doi: 10.1186/1745-6215-15-347. PMID 25187436